CLINICAL TRIAL: NCT05767697
Title: Explore the Correlation of Genomics and Prognosis in Alimentary Tract Cancers
Brief Title: Genomics and Prognosis in GI Cancers
Status: Recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-109-073
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: GI Cancer; Liver Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Clinical biospecimen including blood, plasma, bile, stool, urine, fluid aspirate and tumor/normal tissue will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to collect biospecimens and explore the correlation of genomics and prognosis in alimentary tract cancers.

DETAILED DESCRIPTION:
In this study, the investigators will collect clinical specimens of alimentary tract cancers and perform DNA and RNA analysis to identify genetic alterations for the development of a comprehensive somatic mutation databases and investigate their potential correlation with clinical, radiological and pathological variables. The genomics study included but not limited to target gene panel sequencing, whole exome sequencing, whole genome sequencing, bulk RNA sequencing, single cell RNA sequencing and metagenomics.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign the informed consent
* Age >= 20
* Histology proved pancreatic cancer, esophageal cancer, gastric cancer, hepatocellular carcinoma, cholangiocarcinoma, colorectal cancer
* Agree to provide tumor/normal tissue including but not limited to surgical specimen, biopsy, cytology specimen, bile, urine or stool
* Agree to receive blood sampling 20ml at first time and 10ml during each follow-up (total sampling amount no more than 30ml per month)

Exclusion Criteria:

* Cannot cooperate with blood sampling

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Histology proved pancreatic cancer, esophageal cancer, gastric cancer, hepatocellular carcinoma, cholangiocarcinoma, colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who still survive at 1 year | 1 year
  1 year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, MD PhD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (2):
- Taiwan (2):
  - National Cheng-Kung University Hospital, Tainan
  - National Institute of Cancer Research, Tainan

IPD SHARING:
Plan to Share IPD: No